CLINICAL TRIAL: NCT06222723
Title: Safety and Tolerability of Adjunct Dexamethasone in Addition to Standard of Care Antiviral Therapy Compared to Standard of Care Antiviral Therapy Alone for the Treatment of Moderate to Severe Lassa Fever
Brief Title: LAssa Fever Adjunct Treatment With DEXamethasone
Acronym: LADEX
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bernhard Nocht Institute for Tropical Medicine (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.0 (17 July 2023); 20231908/486 (Other: ISTH EC, Nigeria); 2023-101164-BO-ff (Other: EC Hamburg, Germany)
Record Dates: First submitted 2023-09-29; First posted 2024-01-25 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Lassa Fever
MeSH Terms: conditions — Lassa Fever | interventions — Dexamethasone; Ribavirin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): Standard of care antiviral ribavirin therapy
  Interventions: Drug: Ribavirin
- Standard of care + dexamethasone (Experimental): Standard of care antiviral ribavirin therapy + dexamethasone
  Interventions: Drug: Dexamethasone; Drug: Ribavirin

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone will be administered for 10 days. For the first 48 hours, dexamethasone will be given iv. After 48 hours, a switch to oral dexamethasone (same dosage) is permitted at the discretion of the study physician.
  Arms: Standard of care + dexamethasone
Drug: Ribavirin — Ribavirin treatment will be administered iv for 10 days, as recommended in the Nigeria Centre for Disease Control and Prevention National Guidelines for LF Case Management.

SUMMARY:
Dexamethasone is a corticosteroid which can modulate inflammatory-mediated tissue damage associated with a wide range of infectious diseases. Dexamethasone is routinely used for treatment of tuberculous meningitis and for pneumococcal meningitis in adults. In Coronavirus Disease 2019 (COVID-19) dexamethasone is also effectively preventing immune mediated damage of the lungs. There is also indication that dexamethasone may be promising in severe LF.

DETAILED DESCRIPTION:
Lassa fever (LF) is a severe and often fatal systemic disease in humans. It is caused by the Lassa virus (LASV). Vaccines are not available yet and treatment options are limited to supportive care and ribavirin. Recent LF outbreaks in Nigeria showed an exceptionally high and increasing incidence of LF cases LF affects a large number of countries in West Africa. The pathophysiology of LF is not fully understood yet. It is hypothesized that the damage mediated by the host's defence is plays a key role in the pathophysiology of severe LF. Dexamethasone is considered to dampen the overactive immune response in a range of infectious diseases and thus preventing consecutive damage mediated by the host's immune system, while the antiinfective therapy is effectively treating the underlying pathogen. At the Irrua Specialist Teaching Hospital (ISTH) in Nigeria, one of the largest treatment centres for LF in West-Africa, dexamethasone has been successfully used in clinical practice to manage co-infections of LASV and Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2).

To evaluate Dexamethasone for the treatment of moderate to severe LF cases, a prospective open label randomized controlled phase II clinical trial will be conducted:

1. Standard of care antiviral ribavirin therapy
2. Standard of care antiviral ribavirin therapy + dexamethasone

The primary objective is to assess safety and tolerability of dexamethasone in moderate to severe LF when administered as adjunct treatment. Secondary objectives are to assess the effect of the study intervention on disease progression; to assess immunological and virological impact of dexamethasone therapy and the characterization of population pharmacokinetic characteristics for patients treated with adjunct dexamethasone therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* LF confirmed by RT-PCR (reverse-transcription polymerase chain reaction) with a cycle threshold (Ct) value < 30
* Signs of significant health impairment as evidenced by any of the following:
* Alert, confusion, voice, pain, unresponsive (ACVPU) other than A
* Systolic blood pressure < 90 mmHg
* Seizure(s), meningism, coma, focal neurological deficit
* AST (GOT) >3xULN
* ALT (GPT) > 3xULN
* KDIGO 2 or more severe based on serum creatinine only
* Active macroscopic bleeding
* O2 saturation < 92

Exclusion Criteria:

* Pregnancy (evidenced by positive urine pregnancy test in women of child-bearing potential)
* Lactation following live birth
* Known intolerance and contra-indications to ribavirin or dexamethasone
* Patients who already received a corticosteroid within the preceding 7 days
* Investigator's valuation that patient might be put to substantial risk by participating in this trial
* Patients receiving end-of-life care as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of treatment emergent adverse events and treatment emergent serious adverse events | Participants will be followed up until day 10 after enrollment.
  Documentation of events

SECONDARY OUTCOMES:
Unfavourable outcome | Participants will be followed up until day 10 after enrollment.
  The outcome is measured by the proportion of participants reaching a composite endpoint.
  The outcome is reached if there is a new onset of any of the following: acute kidney injury (KDIGO 3), acute respiratory distress syndrome (SpO2/FiO2 ≤ 315), shock (mean blood pressure < 65 mmHg or systolic blood pressure < 90 mmHg ), encephalopathy (CVPU or seizure), death (yes/no);
Mean/median decline and area under the curve (AUC) of AST, ALT, CK, LDH and CRP | Participants will be followed up until day 10 after enrollment.
  Blood analyses
Description of: proinflammatory plasma cytokine levels and lymphocyte phenotype under treatment | Participants will be followed up until day 10 after enrollment.
  Assays such as the enzyme-linked immunosorbent assays (ELISA) and/or immunofluorescence assays will be used to retrospectively determine LASV IgM and IgG, as well as further IgG subclassification if needed, and to monitor the development of LASV specific antibodies in blood.
  Longitudinal development of inflammatory biomarkers such as IFNα, TNFα, IL-6, and IL-8 will be measured in plasma using bead-based multiplex assays. The phenotype of lymphocytes will be described using flow cytometry.
Description of evolution of viral loads and infectious titers over time until day 10 | Participants will be followed up until day 10 after enrollment.
  Virus titers will be determined. Viral growth, isolation of LASV in cell culture, virus sequencing and unbiased metagenomic sequencing will be used on selected samples to study the longitudinal impact of drug treatment (ribavirin and dexamethasone) on LASV genomes.
Evolution of selected virus gene sequences under treatment | Participants will be followed up until day 10 after enrollment.
  Virus sequencing
Peak plasma concentration (Cmax) | Participants will be followed up until day 10 after enrollment.
  Compartmental analysis
Time to peak plasma concentration (Tmax) | Participants will be followed up until day 10 after enrollment.
  Compartmental analysis
Area under the plasma concentration versus time curve (AUC) | Participants will be followed up until day 10 after enrollment.
  Compartmental analysis
Half life (T 1/2) | Participants will be followed up until day 10 after enrollment.
  Compartmental analysis
Volume of distribution (Vd) | Participants will be followed up until day 10 after enrollment.
  Compartmental analysis

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Günther, Prof., Study Director — Bernhard Nocht Institute for Tropical Medicine
Locations (1):
- Irrua Specialist Teaching Hospital, Irrua, Edo, Nigeria

IPD SHARING:
Plan to Share IPD: No
Case by case decision upon request